CLINICAL TRIAL: NCT06480331
Title: A Randomized Controlled Study on the Efficacy of Ultrasound-guided Fistuloplasty in Comparison to Fluoroscopy-guided Fistuloplasty in Patients With Arteriovenous Access Flow Dysfunction
Brief Title: Radiation Free Fistuloplasty is the Way Forward
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR ID-23-01273-4HI
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-05

CONDITIONS: Fistulas Arteriovenous
Keywords: Endovascular treatments; Percutaneous; Ultrasound
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided fistuloplasty (Experimental): After cleaning and draping the area of interest, local anaesthesia is given to the puncture site. A puncture needle is used to gain access to the arteriovenous fistula followed by a guide wire. Then, a sheath with an appropriate size is placed and a balloon catheter of adequate size is inserted over the guide wire and inflated for 2 minutes. Ultrasound is used in the subject group to monitor technical success. On table visualization of continuous segment of dilated vein to 5-6mm and continuous flow rate of more than 500ml/min signifies the end points of the procedure. After a satisfactory result, a figure of 8 suture is placed with manual inflow occlusion. Post procedure, patients will be observed for any signs of haematoma or bleeding. If there are no immediate complications, patients will be discharged on the same day.
  Interventions: Procedure: Ultrasound-guided fistuloplasty
- Fluoroscopy-guided fistuloplasty (Active Comparator): After cleaning and draping the area of interest, local anaesthesia is given to the puncture site. A puncture needle is used to gain access to the arteriovenous fistula followed by a guide wire. Then, a sheath with an appropriate size is placed and a balloon catheter of adequate size is inserted over the guide wire and inflated for 2 minutes. Ultrasound is used in the subject group to monitor technical success. On table fistulogram visualization of less than 30% recoil of the target lesion signifies technical success. After a satisfactory result, a figure of 8 suture is placed with manual inflow occlusion. Post procedure, patients will be observed for any signs of haematoma or bleeding. If there are no immediate complications, patients will be discharged on the same day.
  Interventions: Procedure: Fluoroscopy-guided fistuloplasty

INTERVENTIONS:
Procedure: Ultrasound-guided fistuloplasty — Radiation free fistuloplasty
  Arms: Ultrasound-guided fistuloplasty
Procedure: Fluoroscopy-guided fistuloplasty — Conventional fistuloplasty
  Arms: Fluoroscopy-guided fistuloplasty

SUMMARY:
The goal of this clinical trial is to study effectiveness of ultrasound-guided fistuloplasty in comparison to conventional fistuloplasty in patients with arteriovenous access flow dysfunction. The main question it aims to answer is:

To investigate patencies in patients with arteriovenous access flow dysfunction receiving ultrasound-guided fistuloplasty versus fluoroscopy-guided fistuloplasty at 6 months

Participants will:

* be randomized equally to ultrasound-guided fistuloplasty group and fluoroscopy-guided fistuloplasty group.
* visit clinic at one month, three month & six months for checkups and tests.

DETAILED DESCRIPTION:
This is an experimental study employing a prospective randomized controlled trial to determine the efficacy of ultrasound-guided fistuloplasty compared to fluoroscopy-guided fistuloplasty in patients with arteriovenous access flow dysfunction.

After assessing for eligibility, patients will be randomized equally with a ratio 1:1 to ultrasound-guided fistuloplasty group and fluoroscopy-guided fistuloplasty group.

Both interventions will be done in operation theatre to maintain sterility. After cleaning and draping the area of interest, local anaesthesia is given to the puncture site. A puncture needle is used to gain access to the arteriovenous fistula followed by a guide wire. Then, a sheath with an appropriate size is placed and a balloon catheter of adequate size is inserted over the guide wire and inflated for 2 minutes. Ultrasound is used in the subject group to monitor technical success. On table visualization of continuous segment of dilated vein to 5-6mm and continuous flow rate of more than 500ml/min signifies the end points of the procedure. Fluoroscopy is used in the control group to assess for technical success. On table fistulogram visualization of less than 30% recoil of the target lesion signifies technical success. After a satisfactory result, a figure of 8 suture is placed with manual inflow occlusion. Post procedure, patients will be observed for any signs of haematoma or bleeding. If there are no immediate complications, patients will be discharged on the same day.

ELIGIBILITY:
Inclusion Criteria:

1. Patient able to comprehend English or Malay language.
2. Patient aged ⩾18 years and ⩽80 years.
3. Patient is willing to comply with protocol.
4. Native AVF that is able to provide prescribed dialysis consistently with 2 needles for >2/3 of dialysis sessions within 4 consecutive weeks.
5. Patient has a reasonable expectation of remaining on haemodialysis for 6 months.
6. Dampened thrill or pulsatile flow.
7. Volume flow (VF) <500 ml/min.
8. Severe stenosis (>50%) of arteriovenous (AV) access measured on color image and confirmed by peak systolic velocity (PSV) ratio of ≥3 in the inflow artery, anastomosis, or in the outflow vein.

Exclusion Criteria:

1. Prior history of fistuloplasty.
2. Thrombosed or completely occluded fistula or outflow vein.
3. Non-mature AVF.
4. Arteriovenous grafts.
5. Suspected central vein stenosis/ cephalic arch stenosis - arm edema or Doppler detected suspicion of the same.
6. Non consenting patient.
7. Metastatic cancer or terminal medical condition.
8. Limited life expectancy (<6 months).
9. Blood coagulation disorders (haemophilia/ Von Willebrand disease/ clotting factor deficiencies/ liver disease).
10. Connective tissue disease (rheumatoid arthritis/ lupus).
11. Sepsis or active infection.
12. Planned access abandonment within 6 months (eg, peritoneal dialysis or transplant).
13. Pregnant women or women of childbearing potential who are not following an effective method of contraception.
14. Allergy or other known contraindication to iodinated media contrast.
15. Patient enrolled in another access maintenance trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To investigate patencies in patients with arteriovenous access flow dysfunction receiving ultrasound-guided fistuloplasty versus fluoroscopy-guided fistuloplasty at 6 months | 6 months
  The duration of time from intervention to thrombosis or any re-intervention to facilitate, maintain, or re-establish patency

SECONDARY OUTCOMES:
To capture data regarding variables that may affect patency of arteriovenous access flow dysfunction post ultrasound-guided fistuloplasty versus fluoroscopy-guided fistuloplasty | Over the course of six months follow-up
  These includes demographic data (comorbidities, smoking history, gender, patient's age, age of fistula) and anatomic location of lesion and number of lesion.
To compare technical success in patients with arteriovenous access flow dysfunction receiving ultrasound-guided fistuloplasty versus fluoroscopy-guided fistuloplasty | Immediately post operation
  Technical success is defined as clinical palpable thrill, radiographic finding of less than 30% recoil and ultrasonographic finding of continuous segment of dilated vein to 5-6mm and continuous flow rate of more than 500ml/min
To compare complication rates in patients with arteriovenous access flow dysfunction receiving ultrasound-guided fistuloplasty versus fluoroscopy-guided fistuloplasty | Immediately post operation
  This includes thrombosis, pseudoaneurysm and bleeding

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Kuala Lumpur Hospital, Jalan Pahang,, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Jln Profesor Diraja Ungku Aziz, Seksyen 13,, Petaling Jaya, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Results will be published by the investigators in academic journals. Sharing of generated study data will be carried out in several different ways. We plan to make our results available to researchers and potential collaborators interested in ultrasound guided fistuloplasty.

REFERENCES:
- [Background] Pisoni RL, Arrington CJ, Albert JM, Ethier J, Kimata N, Krishnan M, Rayner HC, Saito A, Sands JJ, Saran R, Gillespie B, Wolfe RA, Port FK. Facility hemodialysis vascular access use and mortality in countries participating in DOPPS: an instrumental variable analysis. Am J Kidney Dis. 2009 Mar;53(3):475-91. doi: 10.1053/j.ajkd.2008.10.043. Epub 2009 Jan 15. PMID 19150158
- [Background] Tordoir JH, de Bruin HG, Hoeneveld H, Eikelboom BC, Kitslaar PJ. Duplex ultrasound scanning in the assessment of arteriovenous fistulas created for hemodialysis access: comparison with digital subtraction angiography. J Vasc Surg. 1989 Aug;10(2):122-8. doi: 10.1067/mva.1989.0100122. PMID 2668564
- [Background] Leskovar B, Furlan T, Poznic S, Potisek M, Adamlje A, Kljucevsek T. Ultrasound-guided percutaneous endovascular treatment of arteriovenous fistula/graft. Clin Nephrol. 2017 Supplement 1;88(13):61-64. doi: 10.5414/CNP88FX15. PMID 28655388
- [Background] Cho S, Lee YJ, Kim SR. Clinical experience with ultrasound guided angioplasty for vascular access. Kidney Res Clin Pract. 2017 Mar;36(1):79-85. doi: 10.23876/j.krcp.2017.36.1.79. Epub 2017 Mar 31. PMID 28393000
- [Background] Wakabayashi M, Hanada S, Nakano H, Wakabayashi T. Ultrasound-guided endovascular treatment for vascular access malfunction: results in 4896 cases. J Vasc Access. 2013 Jul-Sep;14(3):225-30. doi: 10.5301/jva.5000126. Epub 2013 Jan 8. PMID 23334852
- [Background] Gorin DR, Perrino L, Potter DM, Ali TZ. Ultrasound-guided angioplasty of autogenous arteriovenous fistulas in the office setting. J Vasc Surg. 2012 Jun;55(6):1701-5. doi: 10.1016/j.jvs.2011.12.016. Epub 2012 Jan 23. PMID 22265799
- [Background] Ascher E, Hingorani A, Marks N. Duplex-guided balloon angioplasty of failing or nonmaturing arterio-venous fistulae for hemodialysis: a new office-based procedure. J Vasc Surg. 2009 Sep;50(3):594-9. doi: 10.1016/j.jvs.2009.03.061. PMID 19595550
- [Background] Marks N, Hingorani A, Ascher E. New office-based vascular interventions. Perspect Vasc Surg Endovasc Ther. 2008 Dec;20(4):340-5. doi: 10.1177/1531003508327921. Epub 2008 Nov 19. PMID 19022786
- [Background] Marks N, Ascher E, Hingorani AP. Duplex-guided repair of failing or nonmaturing arterio-venous access for hemodialysis. Perspect Vasc Surg Endovasc Ther. 2007 Mar;19(1):50-5. doi: 10.1177/1531003506298144. PMID 17437980
- [Background] Bacchini G, Cappello A, La Milia V, Andrulli S, Locatelli F. Color doppler ultrasonography imaging to guide transluminal angioplasty of venous stenosis. Kidney Int. 2000 Oct;58(4):1810-3. doi: 10.1046/j.1523-1755.2000.00344.x. PMID 11012917
- [Background] Karmota AG. Paclitaxel coated-balloon (PCB) versus standard plain old balloon (POB) fistuloplasty for failing dialysis access. Ann R Coll Surg Engl. 2020 Oct;102(8):601-605. doi: 10.1308/rcsann.2020.0121. Epub 2020 Jun 15. PMID 32538115
- [Background] Fox D, Amador F, Clarke D, Velez M, Cruz J, Labropoulos N, Ryan M, Gelman L. Duplex guided dialysis access interventions can be performed safely in the office setting: techniques and early results. Eur J Vasc Endovasc Surg. 2011 Dec;42(6):833-41. doi: 10.1016/j.ejvs.2011.04.020. Epub 2011 May 4. PMID 21531585
- [Background] Wittenberg G, Kellner M, Kenn W, Obert A, Schultz G, Trusen A, Tschammler A, Gotz R, Hahn D. [Initial experiences with dilatation of dialysis shunts with color-coded duplex ultrasonography monitoring]. Rofo. 1996 Jan;164(1):38-41. doi: 10.1055/s-2007-1015605. German. PMID 8630358
- See also: Ghanwat SP, Yeramsetti S, Sahu T, Sheorain V, Grover T, Parakh R et al. — http://journals.lww.com/ijvs/fulltext/2021/08010/a_prospective_observational_study_to_evaluate.14.aspx
- See also: Banerjee S, Patel HM, Sahu T, Sheorain VK, Grover T, Parakh R et al. — https://journals.lww.com/ijvs/fulltext/2017/04020/ultrasound_guided_fistuloplasty__a_novel.9.aspx
- See also: Kim JC, Cho JS et al. — https://www.e-ultrasonography.org/journal/view.php?number=507&utm_source=TrendMD&utm_medium=cpc&utm_campaign=Ultrasonography_TrendMD_0

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT06480331/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT06480331/ICF_001.pdf